CLINICAL TRIAL: NCT01039831
Title: The Role of White Matter Pathology in the Development of the Postural Instability and Gait Disturbance (PIGD) Type of Parkinson's Disease (PD)
Brief Title: White Matter Pathology in Parkinson's Disease (PD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Nir Giladi MD, Tel Aviv Sourasky Medical Center
Other Study IDs: 0595-09-TLV
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2009-12

CONDITIONS: White Matter Lesions; Postural Instability Gait Disorders
Keywords: PIGD; tremor; falls; white matter
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Parkinson's Disease: Consecutive patient sampling

SUMMARY:
The relationship between WM lesions (WM) and Postural Instability Gait Disorders (PIGD-PD)in Parkinson's disease patients is largely unknown. We hypothesize that sub-clinical WM pathology may be a major contributing factor to PIGD-PD. We will compare two groups of patients with Parkinson's disease (PD): those with PIGD and patients with dominant tremor (n=120)to assess the role of brain WM changes.

DETAILED DESCRIPTION:
To compare brain WM burden using MRI in PD patients with and without PIGD. Diffusion tensor imaging (DTI) analysis techniques will be applied.We will quantify PIGD-related symptoms including cognitive function, balance and gait and their associations with MRI findings.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD, as defined by the UK Brain Bank criteria
2. Age between 50 and 80 years
3. Hoehn and Yahr stage II-III
4. On anti-parkinsonian medications
5. Mini-Mental State Exam score ≥ 25

Exclusion Criteria:

1. Brain surgery in the past including implanted Deep Brain Stimulation
2. Clinically significant co-morbidities likely to affect gait e.g., acute illness, significant rheumatic, orthopedic disease, dementia, or major depression
3. Unable to walk independently
4. Inability to comply with the protocol

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 120 patients with idiopathic Parkinson's disease (PD) will be studied. Subjects will be divided into two groups: Patients with PIGD and patients with tremor dominant.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, MD, Principal Investigator — Director of the Neurology Department, Tel Aviv Sourasky Medical Center, Israel
Locations (1):
- Laboratory for Gait and Neurodynamics, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel